CLINICAL TRIAL: NCT02236832
Title: Organisation du Cortex préfrontal ventrolatéral Pour l'Analogie: Approche Bimodale Chez le Sujet Sain et Chez le Patient Ayant un Syndrome Frontal.
Brief Title: Study of the Neural Basis of Analogical Reasoning
Acronym: ANALOG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Fondation pour la Recherche Médicale (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: C14-17'; 140662B-31 (Other: ANSM (Agence Nationale de Sécurité du Médicament)); 2014-A00649-38 (Other: ANSM ID RCB)
Record Dates: First submitted 2014-08-28; First posted 2014-09-11 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2017-03

CONDITIONS: Frontotemporal Dementia; Progressive Supranuclear Palsy; Healthy Subjects
MeSH Terms: conditions — Frontotemporal Dementia; Supranuclear Palsy, Progressive | interventions — Transcranial Magnetic Stimulation; Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (5):
- FTD (frontotemporal dementia) patients (Experimental): fronto-temporal demential patients
  Interventions: Other: MRI imaging; Other: EEG recording; Behavioral: Neuropsychological examination
- PSP patients (Experimental): progressive supra nuclear palsy patients
  Interventions: Other: MRI imaging; Other: EEG recording; Behavioral: Neuropsychological examination
- healthy controls (Active Comparator): healthy control education matched, age matched and sex matched with PSP and FTD patients
  Interventions: Other: MRI imaging; Other: EEG recording; Behavioral: Neuropsychological examination
- healthy participants (Experimental): healthy participants that will participate to the TMS study.
  Interventions: Device: transcranial magnetic stimulation; Other: MRI imaging; Other: EEG recording; Behavioral: Neuropsychological examination
- healthy young participants (Experimental): Healthy participants will be included for an EEG study
  Interventions: Other: EEG recording; Behavioral: Neuropsychological examination

INTERVENTIONS:
Device: transcranial magnetic stimulation
  Arms: healthy participants
Other: MRI imaging
  Arms: FTD (frontotemporal dementia) patients; PSP patients; healthy controls; healthy participants
Other: EEG recording
Behavioral: Neuropsychological examination

SUMMARY:
Frontal patients are impaired in categorisation and analogical reasoning tasks, and different functional imaging studies from our group have shown the involvement of the prefrontal cortex in categorisation and analogy tasks. The aim of this project is to test our hypotheses about the role of the prefrontal cortex in explicit and implicit categorisation and analogy tasks.

ELIGIBILITY:
Inclusion Criteria:

Healthy subjects:

* subject affiliated to national health insurance
* informed consent signed
* normal neurological examination
* subject aged at least 20

Patients:

* FTD or PSP diagnostic criteria filled
* patient affiliated to national health insurance
* informed consent signed

Exclusion Criteria:

* Severe psychiatric symptomatology and psychotropic drug use
* unability to understand or perform the cognitive tasks.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2021-02 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
Performance in the implicat task | day of inclusion (one day)
  Reaction time and accuracy will be registered for this categorization task. This task will be used in patients with FTD and in healthy controls (n=60).
  Participants will come only once during one day ot the research centre.
Performance in the Similitude task | from inclusion to 4 months after inclusion
  Reaction time and accuracy will be recorded while healthy subjects perform this categorization task, after a session of rTMS or during on line TMS (n=40).
  Participants will come 3 to 5 times at the research centre in a maximum period of 4 months.

SECONDARY OUTCOMES:
recording of EEG | day of inclusion (one day)
  EEG will be recorded in patients with FTD and in healthy controls for an analysis of event related potentials.
  Participants will come only once during one day a the research centre.
Analysis of MRI | day of inclusion (one day)
  T1 MRI will be recorded for VBM analysis in patients with FTD and healthy controls.
  Participants will come only once during one day at the research centre

CONTACTS AND LOCATIONS:
Overall Officials: Richard Levy, MD, PhD, Principal Investigator — Institut du Cerveau et de la Moelle épinière, Paris
Locations (1):
- ICM (Institut du cerveau et de la Moelle épinière), Paris, France

IPD SHARING:
Plan to Share IPD: Undecided
IPD sharing will be only performed on individual request for a specified study.

REFERENCES:
- [Background] Ovando-Tellez M, Rohaut B, George N, Bieth T, Hugueville L, Ibrahim Y, Courbet O, Naccache L, Levy R, Garcin B, Volle E. Does adding <i>beer</i> to <i>coffee</i> enhance the activation of <i>drinks</i>? An ERP study of semantic category priming. Cogn Neurosci. 2022 Jan-Jun;13(2):61-76. doi: 10.1080/17588928.2021.1940117. Epub 2021 Jul 7. PMID 34232829